CLINICAL TRIAL: NCT04628013
Title: Influence of Noxious Electrical Stimulation on Chronic Pain
Brief Title: Influence of Noxious Electrical Stimulation on Chronic Pain From Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 052820-16
Record Dates: First submitted 2020-10-23; First posted 2020-11-13 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
Keywords: electrical stimulation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The investigators propose a single arm/pre-post trial to examine the effects of NxES on resting pain (BPI, ICOAP), pain sensitivity (PPT, HTS, CPM), movement-related pain (5xSTS), and physical function (5xSTS, KOOS) for people with knee OA. The investigators plan to examine the potential time-course effects after a single intervention (immediate, 1-hr, 24-, and 72-hours) and due to repeated treatment (3x/week for 2-weeks) at the end of treatment (post 72-hours and 4-weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Noxious Electrical Stimulation (NxES) (Experimental): The NxES intervention will be applied for a single treatment in Aim 1 and after a washout period, will be applied 3x/week for 2-weeks (6 sessions) for Aim 2.
  Interventions: Device: Noxious Electrical Stimulation (NxES)

INTERVENTIONS:
Device: Noxious Electrical Stimulation (NxES) — The NxES intervention will be applied with a pair of 2x3 inch electrodes placed orthogonally to the knee joint line with one electrode on the medial and lateral sides of the knee. The device is a commercially available unit(Chattanooga Continuum, DJO Global, Vista CA) and the parameters of the NxES include: 400 μs biphasic square wave pulses delivered at 50-100 pulses/second, using a cycle time of 10-seconds on, with a 2-second ramp-up in intensity, followed by a 10-second off period. The current intensity will be dosed over the first 2-minutes of stimulation to find the sensory perception threshold and the threshold for the first perception of a sharp, prickly buzzing sensation that they would identify as painful. Next, the current intensity will gradually be increased until the participant reports a sharp or prickly buzzing sensation that achieves a pain rating of not more than a 5/10 using a numeric pain rating scale.

SUMMARY:
Knee osteoarthritis (OA) is the most common lower extremity joint pain condition, and it is estimated that 15 million people in the US are living with symptomatic knee OA and that more than half (8 million) are under 65 years of age. To that end, the Centers for Disease Control and Prevention strongly recommends non-pharmacological treatments for chronic pain including physical therapy and weight loss; however, these interventions have significant barriers that can prevent their success. An intervention that targets pain specifically is transcutaneous electrical nerve stimulation (TENS), which is a low-cost intervention with evidence to support pain reduction. As used in the majority of research to date, the intervention called "TENS" refers to the application of electricity across the skin that produces a tingling sensation that is strong but comfortable. However, electricity is applied at a noxious level is thought to result in strong activation of the endogenous pain modulation system, thus producing longer-lasting pain inhibition. However, noxious electrical stimulation (NxES) has rarely been investigated as a treatment intervention. Recent studies, including our own, demonstrate that NxES produces immediate and potentially greater pain relief. Despite some promising research, the clinical use of NxES is sparse and more research is necessary to demonstrate its effects on resting pain, movement-related pain, physical function, and quality of life. The investigators hypothesize that the application of NxES will activate pain modulation mechanisms and change the pain modulation profile toward an anti-nociceptive state in adults with chronic knee osteoarthritis (OA) pain, and thereby decrease pain (at rest and with movement), improve physical function, and improve quality of life. The investigators expect individual differences; therefore, participants will be classified at baseline and their response to the intervention tracked using psychophysical tests and clinical response. The hypothesis will be tested through 2 Specific Aims.

Aim 1: The investigators will test the magnitude and duration of pain relief and functional improvement of a single treatment with NxES in adults with chronic knee OA pain.

Aim 2: The investigators will determine if repeated NxES treatments show greater pain relief and/or functional improvements and if so, whether the gains plateau after a certain number of treatments.

The knowledge gained by this study will be important to physical therapists and other health care practitioners who treat people with chronic knee osteoarthritic pain. If noxious electrical stimulation is found to be an effective strategy to decrease pain at rest and with movement, it may lead to improved patient care, improved function, and decreased chronic pain in people with knee osteoarthritis.

DETAILED DESCRIPTION:
Up to forty-four participants (22 for Aim 1; 22 for Aim 2) with knee OA will be recruited using advertisements, the Legacy Scholars research registry maintained by UNE's Center of Excellence in Aging and Health, from participants with knee OA previously involved in the investigator's research who indicated their willingness to participate in other studies, and from a local orthopedic surgeon group practice. Potential participants will complete a per-participation survey online or by phone that will be used to determine eligibility based on inclusion/exclusion criteria.

For Aims 1 and 2, eligible individuals will be asked to defer any plan for knee joint injections until after the testing period. Participants will be asked to refrain from taking any pain medications for at least 4 hours prior to testing. After giving informed consent, individuals who have diabetes will undergo sensory testing to confirm that their sensory detection threshold is no lower than the mean (+ 2 standard deviations) of the detection threshold of healthy older adults which is 1.4 g of force applied by a size 4.17 monofilament. This threshold is based on data collected in our laboratory using the 4-2-1- method of steps. If the individual is unable to perceive 1.4 g stimulus s/he will not continue in the study.

Protocol for Aim 1- Data collected for Aim 1 will occur over 4 sessions. The purpose of this aim is to determine the magnitude and duration of the day-to-day effects on clinical pain relief and quantitative sensory tests related to pain after a single NxES treatment.

Session 1: In this session we will gain informed consent, then perform a sensory screen (if necessary), collect demographic data and baseline questionnaire data and familiarize participants with the quantitative sensory testing (QST) procedures and to briefly experience the NxES treatment.

Session 2: During this session, participants will experience a single treatment with NxES and we will assess changes in pain and function and QST measures before and after the treatment. For the NxES Intervention, a pair of 2x3 inch electrodes will be placed on the medial and lateral sides of the knee. Pulses of electrical current (400 µs biphasic square wave pulses delivered at 50-100 pulses/second; 10-seconds on: 10-seconds off) will be applied for 20 minutes. The amplitude of the current will be increased until the participant rates the pain 50/100 on numeric pain rating scale. Pain intensity and unpleasantness will be assessed every two-min. and amplitude will be increased to maintain the 5/10 pain intensity level during the treatment. QST will be performed immediately after the treatment and 1 hour later. One- to two-minute washout periods will be provided between QST test repetitions and a 20-minute washout period will be provided after the NxES treatment and the post-treatment test of conditioned pain modulation.

Sessions 3-4: These sessions will occur 24-hours and 72-hours after session 2 and pain and function along with QST will be performed.

Protocol for Aim 2- The purpose of this aim is to determine if there is a cumulative response to NxES treatment on clinical pain and quantitative sensory tests related to pain. Data collected for Aim 2 will begin at least 1-week after the testing for Aim 1 and take place over a 2-week treatment period. Follow-up testing will take place 72-hours and 4-weeks after the last NxES treatment session.

Session 1: This session will be used to re-collect baseline questionnaire data and re-familiarize participants with procedures if it has been greater than 2-weeks since participation in Aim 1 or if they declined participation in Aim 1.

Session 2: During this session, participants will receive the first NxES treatment and undergo assessment of QST, pain, and function.

Session 3-7: These sessions are NxES treatment sessions. Pain and QST assessment will be collected at the beginning of sessions 3,5 & 7 only.

Session 8: No treatments will be performed; post-treatment assessments will occur at 72 hours after session 7.

Session 9: No treatments will be performed; post-treatment assessments will be completed 4 weeks after session 7.

Sessions 2-7 must be completed within 18 calendar days in order to preserve the fidelity of the intervention dosage.

ELIGIBILITY:
Inclusion Criteria:

* follow instructions given in English
* have chronic knee joint-related pain of at least 6-months duration with a pain rating of at least 30/100 mm (0 = no knee pain, 100 = worst imaginable knee pain) over the last 24-hrs.
* report knee pain of at least 30/100 mm with walking, during sit-to-stand transfers, or during stair use

Exclusion Criteria:

* prior experience with NxES
* knee joint injections in the last 3-months or during the time of study participation
* history of total knee arthroplasty in the involved knee
* history of other surgery during the previous 6-months
* history of fibromyalgia or other chronic pain condition
* history of rheumatoid arthritis or related condition
* history of neurologic disorders
* history of cardiovascular or pulmonary disorders that would prevent the completion of the sit-to-stand test
* physician-diagnosed Raynaud's Syndrome
* history of diabetes with diminished sensation
* history of dementia/cognitive impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain Pressure Threshold (PPT medial tibial plateau) | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  PPT will be measured using a pressure algometer (Wagner Instruments, USA; 1cm-squared rubber tip). Pressure will be applied and participants will indicate when the pressure turns to pain. Two trials from each test site with be averaged and used in the analysis. The change in the values from baseline across time points will be analyzed.
Change in Brief Pain Inventory (BPI) | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  The Brief Pain Inventory (BPI) is a 15-question pain questionnaire that examines pain intensity and interference of pain on general activity, mood, walking, work, relationships, sleep and enjoyment of life. The pain intensity sub-scale is score from 0 to 40 points with higher values indicating greater pain intensity. The pain interference sub-scale is scored from 0 to 70 points with higher values indicating greater pain interference. The change in the values from baseline across time points will be analyzed.
Change in Movement-Related Pain | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  Movement-Related Pain will be assessed with a scale on which participants mark their pain intensity on a 100-mm line with 0= "no knee pain" and 100="worst knee pain imaginable". The pain rating will be used to assess pain during functional testing with the 5-times Sit-to-Stand (5xSTS) and the time taken to complete the test will also be recorded and analyzed. The change in the values from baseline across time points will be analyzed.
Change in Intermittent and Constant Osteoarthritis Pain scale (ICOAP) | Aim 1: Assessed at baseline only. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  The Intermittent and Constant Osteoarthritis Pain scale (ICOAP) scale is an 11-item questionnaire; participants rate their constant and intermittent pain on a 5-point scale based on their pain over the past week. The lowest possible score is 0 and the highest score is 100; greater values indicate increasing amounts of pain. The change in the values from baseline across time points will be analyzed.

SECONDARY OUTCOMES:
Change in Conditioned Pain Modulation (CPM) | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  CPM is a test of central pain inhibition. CPM is the difference in PPT measured before and after a painful "conditioning stimulus" is applied. The conditioning stimulus will be immersion of the non-dominant hand in a cold water bath (6-8°C) for 2-minutes. The PPTs will be measured at the wrist of the dominant arm and at the knee at 30- and 90-seconds of immersion. The change in the values from baseline across time points will be analyzed.
Change in Heat Temporal Summation (HTS) | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  HTS is a test of central pain facilitation. It will be completed using a computer-controlled thermode (TSA-II, Medoc, Israel). First, the thermode applies temperature that increases at a rate of 8°C/second until the participant rates thermal pain to be 20-30/100 on the VAS and that temperature (TVAS30) is recorded. Next, the thermode will deliver 10 heat pulses (at a magnitude that will elicit a VAS pain rating of 30/100) once every 2.5 seconds. Participant will provide a VAS after each pulse and difference between the highest and first VAS will be used in the analysis. The change in the values from baseline across time points will be analyzed.
Change in Pressure Pain Threshold (PPT wrist) | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  PPT at the proximal dorsal wrist will be measured using a pressure algometer (Wagner Instruments, USA; 1cm-squared rubber tip). Pressure will be applied and participants will indicate when the pressure turns to pain. Two trials from each test site with be averaged and used in the analysis. The change in the values from baseline across time points will be analyzed.
Change in Five-Times Sit-to-Stand (5xSTS) Test | Aim 1: Assessed at baseline, immediately post-treatment, 24- and 72-hours post-treatment. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  With arms crossed over their chests, participants will rise from a chair and returned to the seated position as quickly as possible for five repetitions and time will be measured in seconds to complete the test. The change in the values from baseline across time points will be analyzed.
Change in Knee injury and Osteoarthritis Outcome score (KOOS) | Aim 1: Assessed at baseline only. Aim 2: Assessed at baseline, at 72-hours after final intervention, and 4-weeks post-intervention.
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self-reported measure that consists of 5 sub-scales (Pain, other Symptoms, Activities of Daily Living, Sports/Recreation, and knee-related Quality of Life). Each sub-scale score is reported on a 0-100 scale, where a 0 indicates extreme symptoms and 100 indicates no symptoms. The change in the values from baseline across time points will be analyzed.

OTHER OUTCOMES:
Pain Catastrophizing Scale (PCS) | Aim 1: Baseline only Aim 2: Baseline only
  The Pain Catastrophizing Scale (PCS) is a 13-item questionnaire designed to quantify an individual's negative behaviors and thoughts in response to actual or potential pain. The total scale ranges from 0-100, with a higher score indicating a greater degree of negative thoughts and behaviors in response to actual and potential pain.
Pain Sensitivity Questionnaire (PSQ) | Aim 1: Baseline only Aim 2: Baseline only
  The Pain Sensitivity Questionnaire (PSQ) is a 17-item questionnaire that asses a patient's perception to various imagined physical stimuli that may be experience in daily life. The scale runs from 0-10, with a higher score indicating greater sensitivity to painful physical stimuli.
Brief Resiliency Scale (BRS) | Aim 1: Baseline only Aim 2: Baseline only
  BRS is a 6-item questionnaire that assesses an individual's ability to bounce back or recover from stress. The possible score range is from 1 (low resilience) to 5 (high resilience).
Depression Anxiety and Stress Scale (DASS-21) | Aim 1: Baseline only Aim 2: Baseline only
  The DASS-21 is a 21-item questionnaire that assess depression, anxiety, and stress symptoms with each construct consisting of a sub-scale with 7-items. Each sub-scale's scores can range from 0 to 42 points, with higher scores representing increasing degrees of the emotional state of depression, anxiety, or stress.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Stackhouse, PT, PhD, Principal Investigator — University of New England
Locations (1):
- University of New England, Portland, Maine, United States

REFERENCES:
- [Background] Stackhouse SK, Taylor CM, Eckenrode BJ, Stuck E, Davey H. Effects of Noxious Electrical Stimulation and Eccentric Exercise on Pain Sensitivity in Asymptomatic Individuals. PM R. 2016 May;8(5):415-24. doi: 10.1016/j.pmrj.2015.07.009. Epub 2015 Aug 3. PMID 26247163
- [Background] Eckenrode BJ, Stackhouse SK. IMPROVED PRESSURE PAIN THRESHOLDS AND FUNCTION FOLLOWING NOXIOUS ELECTRICAL STIMULATION ON A RUNNER WITH CHRONIC ACHILLES TENDINOPATHY: A CASE REPORT. Int J Sports Phys Ther. 2015 Jun;10(3):354-62. PMID 26075151
- [Background] Eckenrode BJ, Kietrys DM, Stackhouse SK. PAIN SENSITIVITY IN CHRONIC ACHILLES TENDINOPATHY. Int J Sports Phys Ther. 2019 Dec;14(6):945-956. PMID 31803527
- [Background] Defrin R, Ariel E, Peretz C. Segmental noxious versus innocuous electrical stimulation for chronic pain relief and the effect of fading sensation during treatment. Pain. 2005 May;115(1-2):152-60. doi: 10.1016/j.pain.2005.02.018. PMID 15836978

DOCUMENTS (1):
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04628013/ICF_000.pdf